CLINICAL TRIAL: NCT04807920
Title: Intravesical OnabotulinumtoxinA Injection at the Time of Prolapse Surgery for the Treatment of Overactive Bladder Syndrome: a Randomized Controlled Trial
Brief Title: BOTOX® at the Time of Prolapse Surgery for OAB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3-2021
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-03

CONDITIONS: Urinary Bladder, Overactive; Pelvic Organ Prolapse
Keywords: Botulinum Toxins, Type A; Mixed Urinary Incontinence; Urgency urinary incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravesical OnabotulinumtoxinA (Experimental): The treatment group will receive 100 units of BOTOX® reconstituted in 10mL of injectable preservative-free normal saline at the time of cystoscopy. An injection cystoscopy needle will be set to 3mm and used to inject 0.5mL reconstituted OnabotulinumtoxinA at each injection site, approximately 1cm apart along the posterior bladder wall, for a total of 20 injection sites (4 rows of 5 injection sites). This will be the only treatment.
  Interventions: Drug: OnabotulinumtoxinA 100 UNT
- Placebo (Placebo Comparator): Subjects randomized to the placebo group will undergo the same procedure but will only receive 10mL of injectable preservative-free normal saline. This will be the only treatment.
  Interventions: Other: Injectable saline

INTERVENTIONS:
Drug: OnabotulinumtoxinA 100 UNT — Intravesical injection
  Arms: Intravesical OnabotulinumtoxinA
Other: Injectable saline — Intravesical injection
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study will be to assess the efficacy and safety of bladder BOTOX® for overactive bladder symptoms, such as urinary urgency and frequency, given at the time of prolapse surgery.

DETAILED DESCRIPTION:
After being informed about the study and the potential risks, women scheduled for prolapse surgery will be screened for bothersome overactive bladder symptoms. Those that qualify and choose to enroll will be randomized to receive either bladder BOTOX® or a placebo at the time of their surgery. Neither the patient nor the investigators will know if the patient receives BOTOX® or a placebo. Subjects will complete questionnaires and bladder diaries both before and after surgery to determine efficacy and patient satisfaction. Potential adverse events, such as urinary tract infections and urinary retention, will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for prolapse surgery
* Bothersome OAB symptoms determined by a score of >20 on the OAB-q SF
* Willingness to perform clean intermittent catheterization (CIC)
* Ability to follow study instructions and complete required follow up

Exclusion Criteria:

* Contraindications or allergy to Onabotulinumtoxin A
* Intravesical Onabotulinumtoxin A within 3 months of the planned surgery date
* Total body Onabotulinumtoxin A dose of ≥ 400 Units in the 3 months prior to the scheduled surgery date.
* Inability or unwillingness to self-catheterize
* Post-void residual ≥ 200mL
* Neurogenic bladder or other neurological diseases that may cause voiding dysfunction
* Concurrent use of other pharmacological treatment for the treatment of OAB symptoms at the time of prolapse repair surgery.
* Females who are pregnant, think they may be pregnant at the start of the study, planning a pregnancy during the active treatment phase of the study, or who are unwilling or unable to use a reliable form of contraception during the active treatment phase of the study.
* Inability to speak or read English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to postoperative weeks 6 to 12 in Overactive Bladder bother short form (OAB-q SF) questionnaire looking for a decrease of 10 points, which is the minimally important difference. | From baseline (time of enrollment) to 6-12 weeks postoperatively
  The OAB-q SF is a validated 6 item questionnaire that is scored and reported on a 0 to 100 point scale with increasing scores indicating more bother.

SECONDARY OUTCOMES:
Change from baseline to postoperative weeks 6 to 12 in the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire short form (PISQ-12). | From baseline (time of enrollment) to 6-12 weeks postoperatively
  The PISQ-12 is a 12 item validated questionnaire that evaluates sexual function in women with urinary incontinence and/or pelvic organ prolapse. It is reported on a scale of 0-48, with a higher score indicating worse sexual function.
Change from baseline to postoperative weeks 6 to 12 in Patient Global Impression of Severity Scale (PGI-S). | From baseline (time of enrollment) to 6-12 weeks postoperatively
  The PGI-S is a 7 point Likert scale, ranging from 1 to 7, with an increasing score indicating greater severity.
Patient Global Impression of Improvement Scale (PGI-I) at 6 to 12 weeks postoperatively. | At 6-12 weeks postoperatively
  The PGI-I is a 7 point Likert scale, ranging from 1 to 7, with an increasing score indicating less improvement.
Urinary tract infection | From time of treatment to 12 weeks postoperative
  Rate of urinary tract infections based on clinical suspicion and urine culture results
Urinary retention | From 2 weeks postoperatively to 12 weeks postoperatively
  Rate of urinary retention requiring catheterization, defined as a post-void residual of more than 400mL or 200-400mL with symptoms of incomplete bladder emptying.

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abrams P, Andersson KE, Birder L, Brubaker L, Cardozo L, Chapple C, Cottenden A, Davila W, de Ridder D, Dmochowski R, Drake M, Dubeau C, Fry C, Hanno P, Smith JH, Herschorn S, Hosker G, Kelleher C, Koelbl H, Khoury S, Madoff R, Milsom I, Moore K, Newman D, Nitti V, Norton C, Nygaard I, Payne C, Smith A, Staskin D, Tekgul S, Thuroff J, Tubaro A, Vodusek D, Wein A, Wyndaele JJ; Members of Committees; Fourth International Consultation on Incontinence. Fourth International Consultation on Incontinence Recommendations of the International Scientific Committee: Evaluation and treatment of urinary incontinence, pelvic organ prolapse, and fecal incontinence. Neurourol Urodyn. 2010;29(1):213-40. doi: 10.1002/nau.20870. No abstract available. PMID 20025020
- [Result] Eapen RS, Radomski SB. Review of the epidemiology of overactive bladder. Res Rep Urol. 2016 Jun 6;8:71-6. doi: 10.2147/RRU.S102441. eCollection 2016. PMID 27350947
- [Result] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Result] Irwin DE, Milsom I, Hunskaar S, Reilly K, Kopp Z, Herschorn S, Coyne K, Kelleher C, Hampel C, Artibani W, Abrams P. Population-based survey of urinary incontinence, overactive bladder, and other lower urinary tract symptoms in five countries: results of the EPIC study. Eur Urol. 2006 Dec;50(6):1306-14; discussion 1314-5. doi: 10.1016/j.eururo.2006.09.019. Epub 2006 Oct 2. PMID 17049716
- [Result] Melville JL, Katon W, Delaney K, Newton K. Urinary incontinence in US women: a population-based study. Arch Intern Med. 2005 Mar 14;165(5):537-42. doi: 10.1001/archinte.165.5.537. PMID 15767530
- [Result] Coyne KS, Sexton CC, Vats V, Thompson C, Kopp ZS, Milsom I. National community prevalence of overactive bladder in the United States stratified by sex and age. Urology. 2011 May;77(5):1081-7. doi: 10.1016/j.urology.2010.08.039. Epub 2011 Jan 22. PMID 21256571
- [Result] Ganz ML, Smalarz AM, Krupski TL, Anger JT, Hu JC, Wittrup-Jensen KU, Pashos CL. Economic costs of overactive bladder in the United States. Urology. 2010 Mar;75(3):526-32, 532.e1-18. doi: 10.1016/j.urology.2009.06.096. Epub 2009 Dec 29. PMID 20035977
- [Result] Minassian VA, Bazi T, Stewart WF. Clinical epidemiological insights into urinary incontinence. Int Urogynecol J. 2017 May;28(5):687-696. doi: 10.1007/s00192-017-3314-7. Epub 2017 Mar 20. PMID 28321473
- [Result] Sexton CC, Coyne KS, Thompson C, Bavendam T, Chen CI, Markland A. Prevalence and effect on health-related quality of life of overactive bladder in older americans: results from the epidemiology of lower urinary tract symptoms study. J Am Geriatr Soc. 2011 Aug;59(8):1465-70. doi: 10.1111/j.1532-5415.2011.03492.x. Epub 2011 Jun 30. PMID 21718275
- [Result] Lightner DJ, Gomelsky A, Souter L, Vasavada SP. Diagnosis and Treatment of Overactive Bladder (Non-Neurogenic) in Adults: AUA/SUFU Guideline Amendment 2019. J Urol. 2019 Sep;202(3):558-563. doi: 10.1097/JU.0000000000000309. Epub 2019 Aug 8. PMID 31039103
- [Result] Brubaker L, Richter HE, Visco A, Mahajan S, Nygaard I, Braun TM, Barber MD, Menefee S, Schaffer J, Weber AM, Wei J; Pelvic Floor Disorders Network. Refractory idiopathic urge urinary incontinence and botulinum A injection. J Urol. 2008 Jul;180(1):217-22. doi: 10.1016/j.juro.2008.03.028. Epub 2008 May 21. PMID 18499184
- [Result] Chapple C, Sievert KD, MacDiarmid S, Khullar V, Radziszewski P, Nardo C, Thompson C, Zhou J, Haag-Molkenteller C. OnabotulinumtoxinA 100 U significantly improves all idiopathic overactive bladder symptoms and quality of life in patients with overactive bladder and urinary incontinence: a randomised, double-blind, placebo-controlled trial. Eur Urol. 2013 Aug;64(2):249-56. doi: 10.1016/j.eururo.2013.04.001. Epub 2013 Apr 10. PMID 23608668
- [Result] Dmochowski R, Chapple C, Nitti VW, Chancellor M, Everaert K, Thompson C, Daniell G, Zhou J, Haag-Molkenteller C. Efficacy and safety of onabotulinumtoxinA for idiopathic overactive bladder: a double-blind, placebo controlled, randomized, dose ranging trial. J Urol. 2010 Dec;184(6):2416-22. doi: 10.1016/j.juro.2010.08.021. Epub 2010 Oct 16. PMID 20952013
- [Result] Drake MJ, Nitti VW, Ginsberg DA, Brucker BM, Hepp Z, McCool R, Glanville JM, Fleetwood K, James D, Chapple CR. Comparative assessment of the efficacy of onabotulinumtoxinA and oral therapies (anticholinergics and mirabegron) for overactive bladder: a systematic review and network meta-analysis. BJU Int. 2017 Nov;120(5):611-622. doi: 10.1111/bju.13945. Epub 2017 Aug 2. PMID 28670786
- [Result] Fowler CJ, Auerbach S, Ginsberg D, Hale D, Radziszewski P, Rechberger T, Patel VD, Zhou J, Thompson C, Kowalski JW. OnabotulinumtoxinA improves health-related quality of life in patients with urinary incontinence due to idiopathic overactive bladder: a 36-week, double-blind, placebo-controlled, randomized, dose-ranging trial. Eur Urol. 2012 Jul;62(1):148-57. doi: 10.1016/j.eururo.2012.03.005. Epub 2012 Mar 14. PMID 22464310
- [Result] Herschorn S, Kohan A, Aliotta P, McCammon K, Sriram R, Abrams S, Lam W, Everaert K. The Efficacy and Safety of OnabotulinumtoxinA or Solifenacin Compared with Placebo in Solifenacin Naive Patients with Refractory Overactive Bladder: Results from a Multicenter, Randomized, Double-Blind Phase 3b Trial. J Urol. 2017 Jul;198(1):167-175. doi: 10.1016/j.juro.2017.01.069. Epub 2017 Feb 1. PMID 28161352
- [Result] Visco AG, Brubaker L, Richter HE, Nygaard I, Paraiso MF, Menefee SA, Schaffer J, Lowder J, Khandwala S, Sirls L, Spino C, Nolen TL, Wallace D, Meikle SF; Pelvic Floor Disorders Network. Anticholinergic therapy vs. onabotulinumtoxina for urgency urinary incontinence. N Engl J Med. 2012 Nov 8;367(19):1803-13. doi: 10.1056/NEJMoa1208872. Epub 2012 Oct 4. PMID 23036134
- [Result] Sexton CC, Notte SM, Maroulis C, Dmochowski RR, Cardozo L, Subramanian D, Coyne KS. Persistence and adherence in the treatment of overactive bladder syndrome with anticholinergic therapy: a systematic review of the literature. Int J Clin Pract. 2011 May;65(5):567-85. doi: 10.1111/j.1742-1241.2010.02626.x. PMID 21489081
- [Result] Sussman D, Yehoshua A, Kowalski J, Lee W, Kish J, Chaudhari S, Murray B. Adherence and persistence of mirabegron and anticholinergic therapies in patients with overactive bladder: a real-world claims data analysis. Int J Clin Pract. 2017 Mar;71(3-4):e12824. doi: 10.1111/ijcp.12824. PMID 28371019
- [Result] Dmochowski RR, Thai S, Iglay K, Enemchukwu E, Tee S, Varano S, Girman C, Radican L, Mudd PN Jr, Poole C. Increased risk of incident dementia following use of anticholinergic agents: A systematic literature review and meta-analysis. Neurourol Urodyn. 2021 Jan;40(1):28-37. doi: 10.1002/nau.24536. Epub 2020 Oct 23. PMID 33098213
- [Result] Clinical Consensus Statement: Association of Anticholinergic Medication Use and Cognition in Women With Overactive Bladder. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):69-71. doi: 10.1097/SPV.0000000000001008. PMID 33497068
- [Result] Granese R, Adile G, Gugliotta G, Cucinella G, Saitta S, Adile B. Botox((R)) for idiopathic overactive bladder: efficacy, duration and safety. Effectiveness of subsequent injection. Arch Gynecol Obstet. 2012 Oct;286(4):923-9. doi: 10.1007/s00404-012-2349-8. Epub 2012 May 24. PMID 22622849
- [Result] Shepherd JP, Carter-Brooks CM, Chermanksy C. A cost-effectiveness analysis of Onabotulinumtoxin A as first-line treatment for overactive bladder. Int Urogynecol J. 2018 Aug;29(8):1213-1219. doi: 10.1007/s00192-018-3653-z. Epub 2018 Apr 18. PMID 29671033
- [Result] de Boer TA, Salvatore S, Cardozo L, Chapple C, Kelleher C, van Kerrebroeck P, Kirby MG, Koelbl H, Espuna-Pons M, Milsom I, Tubaro A, Wagg A, Vierhout ME. Pelvic organ prolapse and overactive bladder. Neurourol Urodyn. 2010;29(1):30-9. doi: 10.1002/nau.20858. PMID 20025017
- [Result] Johnson JR, High RA, Dziadek O, Ocon A, Muir TW, Xu J, Antosh DD. Overactive Bladder Symptoms After Pelvic Organ Prolapse Repair. Female Pelvic Med Reconstr Surg. 2020 Dec 1;26(12):742-745. doi: 10.1097/SPV.0000000000000700. PMID 30681419
- [Result] de Boer TA, Kluivers KB, Withagen MI, Milani AL, Vierhout ME. Predictive factors for overactive bladder symptoms after pelvic organ prolapse surgery. Int Urogynecol J. 2010 Sep;21(9):1143-9. doi: 10.1007/s00192-010-1152-y. Epub 2010 Apr 24. PMID 20419366
- [Result] Foster RT Sr, Barber MD, Parasio MF, Walters MD, Weidner AC, Amundsen CL. A prospective assessment of overactive bladder symptoms in a cohort of elderly women who underwent transvaginal surgery for advanced pelvic organ prolapse. Am J Obstet Gynecol. 2007 Jul;197(1):82.e1-4. doi: 10.1016/j.ajog.2007.02.049. PMID 17618768
- [Result] Sung VW, Borello-France D, Newman DK, Richter HE, Lukacz ES, Moalli P, Weidner AC, Smith AL, Dunivan G, Ridgeway B, Nguyen JN, Mazloomdoost D, Carper B, Gantz MG; NICHD Pelvic Floor Disorders Network. Effect of Behavioral and Pelvic Floor Muscle Therapy Combined With Surgery vs Surgery Alone on Incontinence Symptoms Among Women With Mixed Urinary Incontinence: The ESTEEM Randomized Clinical Trial. JAMA. 2019 Sep 17;322(11):1066-1076. doi: 10.1001/jama.2019.12467. PMID 31529007
- [Result] Miotla P, Futyma K, Cartwright R, Bogusiewicz M, Skorupska K, Markut-Miotla E, Rechberger T. Effectiveness of botulinum toxin injection in the treatment of de novo OAB symptoms following midurethral sling surgery. Int Urogynecol J. 2016 Mar;27(3):393-8. doi: 10.1007/s00192-015-2839-x. Epub 2015 Sep 12. PMID 26364180
- [Result] Komar A, Bretschneider CE, Mueller MG, Lewicky-Gaupp C, Collins S, Geynisman-Tan J, Tavathia M, Kenton K. Concurrent Retropubic Midurethral Sling and OnabotulinumtoxinA for Mixed Urinary Incontinence: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jan 1;137(1):12-20. doi: 10.1097/AOG.0000000000004198. PMID 33278293